CLINICAL TRIAL: NCT01504802
Title: Pharmacodynamics of C-Type Natriuretic Peptide During Growth Hormone Treatment in Children: A Potential Biomarker of Efficacy
Brief Title: Pharmacodynamics of CNP During Growth Hormone Treatment
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Children's Hospital Los Angeles (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Rob Olney, Physician/Researcher, Nemours Children's Clinic
Other Study IDs: NCC 167624
Record Dates: First submitted 2011-07-20; First posted 2012-01-05 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Pituitary Dwarfism; Idiopathic Short Stature
Keywords: Growth hormone; C-type natriuretic peptide; amino-terminal propeptide of C-type natriuretic peptide; insulin-like growth factor-I; bone specific alkaline phosphatase; leptin; deoxypyridinoline; growth velocity; pharmacodynamic; biomarker
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, and urine will be saved for potential future studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Growth hormone deficient: Children with short stature, a peak growth hormone response on stimulation testing of less than 7 ng/ml, and no other identifiable cause of short stature
- Idiopathic short stature: Children with short stature, a peak growth hormone response on stimulation testing of greater than or equal to 7 ng/ml, and no identifiable cause for the short stature

SUMMARY:
It is now widespread practice to treat children with short stature with growth hormone. However, how an individual child will respond to growth hormone treatment is unpredictable and highly variable. Some children will not respond to growth hormone treatment at all. Currently, the only way to determine how well growth hormone therapy is working is to wait until they have been treated for six months and to compare the pre-treatment growth velocity with the growth velocity on treatment. It would be helpful to have a blood test that could be done shortly after starting growth hormone that could predict whether how well a child is responding to treatment. Such a blood test would allow endocrinologists to adjust the growth hormone dose (or possibly stop it altogether, if it is not working) long before the six months it currently takes.

C-type natriuretic peptide (CNP) and its partner amino-terminal propeptide of CNP (NTproCNP) are proteins that play a critical role in regulating growth. The investigators have previously shown that blood levels of these proteins increase in children being treated with growth hormone. The investigators believe that a blood test for these proteins will be useful in predicting a child's response to growth hormone treatment.

The purpose of this study is to determine when after starting growth hormone, the blood levels of CNP and NTproCNP start to increase.

DETAILED DESCRIPTION:
Treatment of children with short stature with recombinant human growth hormone is widespread practice. However, the growth response to growth hormone treatment is highly variable, particularly for those children who do not have classic growth hormone deficiency. The availability of a biomarker of efficacy that can be measured early in treatment would be beneficial.

C-type natriuretic peptide (CNP) plays a critical role in linear growth. CNP is produced in the growth plate and signals through a paracrine mechanism. Its bioinactive amino-terminal propeptide (NTproCNP) is easily measurable in plasma and levels reflect rate of CNP biosynthesis. Previous studies in lambs and children have shown that the plasma concentration of NTproCNP correlates with linear growth velocity and the investigators have also shown that levels are increased during growth hormone therapy. The investigators have proposed that NTproCNP is a biomarker for linear growth and consider it the first "growth plate function test." Such a growth biomarker is likely to reflect efficacy of growth hormone therapy soon after starting growth hormone, possibly as soon as a few days. Before the clinical utility of this can be determined, the investigators need to ascertain the pharmacodynamics of CNP and NTproCNP in response to growth hormone.

The goal of this study is to describe the pharmacodynamics of the CNP response to the initiation of growth hormone in two sets of children with short stature, those with growth hormone deficiency and those in whom normal growth hormone secretion (idiopathic short stature) and to compare these data to the pharmacodynamics of other peptides previously identified as potential biomarkers. The investigators hypothesize that plasma NTproCNP levels will increase within four days of starting growth hormone therapy and that the response in children with growth hormone deficiency will be more prompt and greater than those with idiopathic short stature. The investigators second hypothesis is that the increase in NTproCNP in response to growth hormone will correlate with the increase in growth velocity after six and twelve months of treatment.

The study is a prospective observational study of children with growth hormone deficiency (n=10) and with idiopathic short stature (n=10) being started on rhGH therapy. The study consists of frequent monitoring of analyte levels over one year of treatment.

This is a two site study, Nemours Children's Clinic, Jacksonville, Florida and Children's Hospital Los Angeles.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 3 years
* Prepubertal
* Height SD score less than -2.25
* Had a growth hormone stimulation test

Exclusion Criteria:

* History of any other disease or drug treatment that might interfere with linear growth, including amphetamine derivatives for treatment of ADD or ADHD
* Previous treatment with any growth-promoting medication, including growth hormone
* Any contraindication to growth hormone therapy
* Minor acute illness (upper respiratory infections, strep throat, gastroenteritis, urinary tract infection, etc.) less than one month prior to starting growth hormone
* Major acute illness (pneumonia, meningitis, pyelonephritis, any illness requiring hospitalization, etc.), any surgery, or bone fracture less than six months prior to starting growth hormone
* Weight less than 13 kg (NCC-J) or 15 kg (CHLA), due to blood volume being drawn.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with short stature
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Determine the time after starting rhGH that NTproCNP level reaches 95% of its peak level | One year
  NTproCNP will be modeled over time for each individual subject and the time it reaches 95% of its peak value determined. This value will then be averaged for the cohort.

SECONDARY OUTCOMES:
Correlate NTproCNP levels at the time it reaches 95% of its peak with six-month and one year growth velocity on rhGH treatment | one year
Compare NTproCNP levels with other biomarkers of growth (serum IGF-I, bone-specific alkaline phosphatase, and leptin, and urine deoxypyridinoline) during rhGH treatment | One year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olney, MD, Principal Investigator — Nemours Children's Clinic
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Nemours Children Clinic, Jacksonville, Florida

REFERENCES:
- See also: Nemours Children's Clinic — http://www.Nemours.org